CLINICAL TRIAL: NCT02098291
Title: Phase II, Open, Single-center Study to Determine the Antibody Response to Gastrimmune and Its Safety and Tolerability in Patients With Advanced Pancreatic Carcinoma
Brief Title: An Open, Single-center Study to Determine the Antibody Repsonse to Gastrimmune and Its Safety and Tolerability in Patients With Advanced Pancreatic Carcinoma
Acronym: PC1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC1
Record Dates: First submitted 2014-03-12; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

ARMS (1):
- G17DT (Experimental)
  Interventions: Drug: G17DT

INTERVENTIONS:
Drug: G17DT

SUMMARY:
This study was designed to determine the effect of jaundice on the ability of G17DT to generate antibodies before and after treatment of biliary obstruction due to advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological confirmation of pancreatic carcinoma who were not suitable for pancreatic tumour resection with curative intent
* Patients who had not received chemotherapy in the previous month and who would either not receive chemotherapy in the period of study or who would commence gemcitabine treatment in week 4 of the study
* Male or female patients over 18 years of age
* Patients with a life expectancy of at least 2 months
* Patients must have given written informed consent
* Patients with a Karnofsky Performance Status score of ≥ 50%
* Patients who would not receive chemotherapy in the period of the Extension Survival Study, except for concomitant gemcitabine ongoing at visit (for extension study)

Exclusion Criteria:

* History of other malignant disease except non-melanomatous skin carcinoma or in situ carcinoma of the uterine cervix
* Concomitant use or anticipated use in the period of the study of radiotherapy
* Chemotherapy in the previous month preceding screening, anticipated concomitant use of chemotherapy between screening and week 4 of the study or anticipated useof chemotherapeutic agents other than gemcitabine from week 4 for the period of the study
* Use in the past month or concomitant use of immunosuppressants, including systemic (i.e. oral or injected) corticosteroids
* Females who were pregnant, planning to become pregnant or lactating
* Patients taking part in another study involving an investigational or licensed drug or device in the three months preceding enrolment or during the study
* Haematological indicators:

Haemoglobin <9.5g/dl White blood cell count <3.5 x 109/l Platelets <100 x 109/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 1999-04; Primary Completion 2001-07 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic | Up to week 16
  Anti-Gastrin 17 antibodies were determined at baseline (week0) and measured at subsequent visits during the first 16 weeks after the first G17DT injection to determine the effect of jaundice on the ability of patients to generate antibodies.

SECONDARY OUTCOMES:
Patient Survival | Up to week 139
  The vital status was monitored throughout the study and was followed up to the death of the last patient.
Number of Participants with Serious and Non-Serious Adverse Events | Up to week 60
  Adverse events, defined as any event involving adverse reactions, illnesses with onset during the study, or exacerbations of pre-exisiting illnesses, were assessed at each visit.